CLINICAL TRIAL: NCT05475067
Title: Fever Tracking Study: The Feasibility of Fever Tracking in a Home-setting by a Non-invasive Wearable Core Body Temperature Sensor
Brief Title: Fever Tracking Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: greenTEG AG (Industry)
Responsible Party: Sponsor
Other Study IDs: Fever Tracking
Record Dates: First submitted 2022-06-01; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Core Body Temperature in Healthy Subjects; Immune Response to mRNA COVID-19 Vaccination
Keywords: Fever Tracking; Core body temperature CBT; mRNA COVID-19 vaccination; Wearable sensors; Wearables

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the feasibility of continuous fever tracking of participants having fever symptoms in a home setting, using a core body temperature (CBT) sensor. CBT as measured by the wearable sensors will be coampared with CBT as measured by ingestible electronc pills (reference).

A secondary research question is, if the CBT behavior of the the participants in a home setting can be compared to previously described CBT profiles in the literature, and if special patterns can be identified.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Informed consent signed
* Either:

Acute fever symptoms at inclusion (at least 38.0°C) and Test for COVID-19 at the day of inclusion

- Or: Second shot or booster of mRNA COVD-19 vaccination (Comirnaty® or COVID-19 Vaccine Moderna®) at day of inclusion

Exclusion Criteria:

* Any participant who, for any reason, is unable to independently consent to participate in the study and/or who is unable to independently follow the study protocol.
* Any participant with previous surgical procedures in the gastrointestinal tract
* Inability to swallow pills
* Any participant of ≤40 kg body weight
* A scheduled MRI examination in the period from the start of the measurements until seven days after ingestion of the electronic pill.
* Any participant being pregnant
* Impairment or disability of the upper extremity likely to have a negative impact on the quality of measurements:

  * Wounds
  * Active venous access
  * Amputations
  * Dialysis shunt
  * Edema
  * Axillary dissection
  * Continuous long-term monitoring of blood pressure
  * Tattoos
* Known allergy to plastics / latex
* Language problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects testing for COVID-19 at the University Hospital Basel and having acute fever symptoms, or individuals receiving the second shot or the booster of an mRNA COVID 19 vaccination, will be informed about the possibility to participate in this study by study personnel on-site.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Mean absolute error, bias and standard deviation of the predicted CBT by the wearable CBT sensor compared to the reference temperature method (ingestible electronic pill) | 48 hours
  This comparison will be done for each position of the wearable CBT sensor (apical, upper arm and wrist).

SECONDARY OUTCOMES:
Mean absolute error, mean bias and standard deviation of the predicted CBT sensor compared to the reference temperature method (ingestible electronic pill). | 48 hours
  In addition to the primary outcome measure, the heartrate will be used as additional input to perform the CBT prediction of the wearables.

OTHER OUTCOMES:
Influence of age on the predicted CBT | 48 hours
  Age measured in years
Influence of sex on the predicted CBT | 48 hours
Influence of weight on the predicted CBT | 48 hours
  Weight measured in kg
Influence of height on the predicten CBT | 48 hours
  Height measured in cm
Influence of skin colour on the predicted CBT | 48 hours
  Skin colour measured on the Fitzpatrick Skin Type Scala which classifies skin types from I to VI, depending on the amount of melanin pigment. Type I contains the lowest level of melanin, whereas type VI has the highest level.
Influence of hairiness on the predicted CBT | 48 hours
  Degree of hairiness expressed as mild, moderate and strong
Influence of food intake on the predicted CBT | 48 hours
  The impact of the above mentioned factor on the CBT will be monitored and recorded in a participant diary
Influence of concomitant medications on the predicted CBT | 48 hours
  The impact of the above mentioned factors on the CBT will be monitored and recorded in a participant diary

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Universitiy Hospital Basel, Basel, Canton of Basel-City, Switzerland